CLINICAL TRIAL: NCT04049695
Title: A Randomized Trial of Physical Activity for Cognitive Functioning in Breast Cancer Survivors
Brief Title: Improving Cognition After Cancer
Acronym: ICAN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sheri Hartman, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 182113
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer Survivors; Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): This arm will receive a 12-month individually tailored phone and email-based exercise program.
  Interventions: Behavioral: Exercise
- Health & Wellness Intervention (Active Comparator): This arm will receive a 12-month health and wellness program.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Exercise — This intervention is based on Control Theory and Social Cognitive Theory and includes: 1) weekly emails with tips and tools to set personalized exercise goals and to increase exercise; 2) Health coaching phone sessions; 3) wrist worn monitor such as a Fitbit to track activity
  Arms: Exercise Intervention
Behavioral: Control — This intervention includes: 1) weekly emails with tips and tools to support health and wellness such as brain health, stress management, nutrition; 2) Health coaching phone sessions
  Arms: Health & Wellness Intervention

SUMMARY:
This study will test whether a physical activity intervention can improve cognition in breast cancer survivors and help the development of physical activity guidelines for cognition in breast cancer survivors.

DETAILED DESCRIPTION:
Many breast cancer survivors experience problems with mental abilities such as memory, attention, and concentration (known as cognition). Increasing physical activity has been shown to improve cognition in adults; however, little is known about whether this is helpful for cancer survivors as well. This study will test whether a physical activity intervention can improve cognition in breast cancer survivors and help the development of physical activity guidelines for cognition in breast cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer survivors who have completed active treatment at least 6 months prior to enrollment and are within 5 years of diagnosis of stage 1, 2, or 3 breast cancer
* self-report difficulties with cognition since their cancer diagnosis
* self-report low levels of moderate to vigorous physical activity
* have a Fitbit compatible device with internet
* breast cancer was treated with chemotherapy and/or hormonal therapy

Exclusion Criteria:

* medical condition that could make it potentially unsafe to be in an unsupervised physical activity intervention
* currently taking tamoxifen or aromatase inhibitor that will be stopped in the next 6 months
* unable to commit to a 12-month study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 253 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
National Institutes of Health Toolbox - Cognition Domain - Oral Symbol Digital Test | Baseline to 6 months
  Measure of processing speed

SECONDARY OUTCOMES:
National Institutes of Health Toolbox - Cognition Domain - Oral Symbol Digital Test | Baseline to 12 months
  Measure of processing speed
Patient Reported Outcomes Measurement Information System (PROMIS) cognitive abilities | Baseline to 6 months and Baseline to 12 months
  Measure of Self-Report Cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Moores UCSD Cancer Center, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT04049695/ICF_000.pdf